CLINICAL TRIAL: NCT03836287
Title: A Multicenter, Randomized, Double-Blinded, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of Topically Applied Sofpironium Bromide Gel, 15% in Subjects With Axillary Hyperhidrosis
Brief Title: Safety and Efficacy Study of Sofpironium Bromide in Subjects With Axillary Hyperhidrosis (BBI-4000-CL-301)
Acronym: CardiganI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Botanix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBI-4000-CL-301
Record Dates: First submitted 2019-02-06; First posted 2019-02-11 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Axillary Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Sofpironium bromide, 15% gel, once per day
  Interventions: Drug: Sofpironium Bromide Gel, 15%
- Vehicle (Placebo Comparator): Vehicle gel, once per day
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Sofpironium Bromide Gel, 15% — Active
  Other Names: BBI-4000 Gel, 15%
  Arms: Active
Drug: Vehicle — Vehicle gel
  Other Names: BBI-4000 Gel, 0%
  Arms: Vehicle

SUMMARY:
Hyperhidrosis is a disorder of abnormal excessive sweating. Primary hyperhidrosis (armpits, hands, and feet) affects approximately 4.8% of the US population and is believed to be caused by an overactive cholinergic response of the sweat glands.

Current therapies have limited effectiveness, significant side effects, and can be invasive and costly. Sofpironium bromide (BBI-4000) is a novel soft-drug in development for the topical treatment of hyperhidrosis.

This Phase 3 study will assess the safety and efficacy of sofpironium bromide, 15% gel versus vehicle (2 treatment arms), applied for the treatment of axillary hyperhidrosis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, vehicle-controlled study to evaluate the safety and efficacy of topically applied sofpironium bromide, 15% gel in subjects with axillary hyperhidrosis.

Safety will be assessed through collection of vital signs, adverse events, local skin responses, hematology, serum chemistry laboratory testing and urinalysis.

A maximum of 350 subjects will be randomized to receive either sofpironium bromide gel, 15% or vehicle.

Adverse events, vital signs, and local tolerability assessments will be collected at visits across the study. Urine pregnancy tests will be taken throughout the course of the study for women of child bearing potential. Blood and urine samples will be collected and analyzed for routine hematology, chemistry, and urinalysis parameters at specified visits. Patient-reported outcome assessments will be recorded during the study at predefined time points.

The study will be comprised of a total of 13 scheduled visits to take place over approximately 11 to 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥ 9 years of age.
* Diagnosis of primary axillary hyperhidrosis that meets the following criteria: (a) symptoms of hyperhidrosis for at least 6 months' duration, (b) HDSM-Ax of 3 - 4 and (c) a minimum GSP of 50 mg in each axilla with a combined total of at least 150 mg.
* The ability to understand and follow all study-related procedures including study drug administration.
* Sexually active female of childbearing potential (FOCBP)* must agree to periodic pregnancy testing and use a medically acceptable method of contraception while receiving protocol-assigned product.

Exclusion Criteria:

* In the Investigators opinion, any skin or subcutaneous tissue conditions of the axilla(e).
* Prior use of any prohibited medication(s) or procedure(s) within the specified timeframe for the treatment of axillary hyperhidrosis.
* Anticholinergic agents used to treat conditions such as, but not limited to, hyperhidrosis, asthma, incontinence, gastrointestinal cramps, and muscular spasms by any route of administration.
* Use of any cholinergic drug (e.g. bethanechol) within 28 days.
* Known cause of hyperhidrosis or known history of a condition that may cause hyperhidrosis (i.e., hyperhidrosis secondary to any known cause such hyperthyroidism, diabetes mellitus, medications, etc.).
* Subjects with unstable diabetes mellitus or thyroid disease, history of renal or hepatic impairment, malignancy glaucoma, intestinal obstructive or motility disease, obstructive uropathy, myasthenia gravis, BPH, neurological or psychiatric conditions, Sjögren's or Sicca syndrome, or cardiac abnormalities that may alter or exacerbate sweat production by the use of anticholinergics in the investigator's opinion.
* Subjects with known hypersensitivity to glycopyrrolate, anticholinergics, or any of the components of the topical formulation.
* Subject is pregnant, lactating or is planning to become pregnant during the study.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walker, MD PhD, Study Director — Botanix Pharmaceuticals
Locations (39):
- United States (39):
  - Total Skin and Beauty Dermatology Center, P.C., Birmingham, Alabama
  - Investigate MD, LLC, Scottsdale, Arizona
  - Northwest Arkansas Clinical Trials Center, Rogers, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Dermatology Research Associates, Los Angeles, California
  - Therapeutics Clinical Research, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - AboutSkin Research, LLC, Greenwood Village, Colorado
  - Center for Clinical & Cosmetic Research, Aventura, Florida
  - Skin Care Research, LLC, Boca Raton, Florida
  - Skin Research Institute, Coral Gables, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - Aby's New Generation Research, Hialeah, Florida
  - Baumann Cosmetic and Research Institute, Miami, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - My Community Research Center, Inc., Miami, Florida
  - Tory Sullivan, MD PA, North Miami Beach, Florida
  - Research Institute of the Southeast, West Palm Beach, Florida
  - Dawes Fretzin Research Group, Indianapolis, Indiana
  - Maryland Laser Skin and Vein, Hunt Valley, Maryland
  - Lawrence J Green, MD LLC, Rockville, Maryland
  - SkinCare Physicians, Chestnut Hill, Massachusetts
  - Grekin Skin Institute, Warren, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Skin Specialists, P.C., Omaha, Nebraska
  - Hassman Research Institute, Berlin, New Jersey
  - DermResearch Center of New York, Inc., Stony Brook, New York
  - PMG Research of Cary, Raleigh, North Carolina
  - Haber Dermatology and Cosmetic Surgery, Inc., Beachwood, Ohio
  - Oregon Dermatology & Research Center, Portland, Oregon
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Dermatology Associates of Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Vehicle
Started | 173 | 177
Completed | 150 | 162
Not Completed | 23 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Vehicle | Total
Number analyzed (Participants) | 173 | 177 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (11.63) | 32.4 (10.86) | 32.7 (11.21)
Age, Customized [Count of Participants; unit: Participants]
  9-12 years | 2 | 0 | 2
  13-16 years | 7 | 9 | 16
  17-30 years | 70 | 73 | 143
  ≥31 years | 94 | 95 | 189
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 99 | 197
  Male | 75 | 78 | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61 | 60 | 121
  Not Hispanic or Latino | 111 | 117 | 228
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 43 | 74
  White | 140 | 130 | 270
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Time Since Start of Axillary Hyperhidrosis Symptoms [Mean (Standard Deviation); unit: Months] | 179.29 (115.155) | 184.42 (116.898) | 181.86 (115.708)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Vehicle Arm vs. Sofpironium Bromide Gel, 15%) With and Without an Observed ≥2-point Improvement in Hyperhidrosis Disease Severity Measure-Axillary-7 Item Total Score From Baseline to End of Treatment
Description: Change in score from baseline to end of treatment of 7 questions from the patient reported outcome assessment - Hyperhidrosis Disease Severity Measure-Axillary-7; each question had a 5-point response (range 0 [better] - 4 [worse]). Total scores were calculated by averaging the score of all items, resulting in an axillary hyperhidrosis symptom range of 0 (no sweating) to 4 (worst possible sweating). Improvement corresponded to a ≥2-point reduction of individual participant score from baseline to end of treatment (end of treatment [6 weeks] score minus baseline score). Treatment arms compared included vehicle and Sofpironium Bromide Gel, 15%. Counts of participants (per treatment arm) with and without an observed ≥2-point improvement in Hyperhidrosis Disease Severity Measure-Axillary-7 Item Total Score from baseline to end of treatment were used as the outcome value(s).
Time Frame: Total Trial Participation was approximately 11-15 weeks; outcome measure time frame: Baseline (and treatment start) through to end of treatment, taking approximately 6 weeks.
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Vehicle
Number analyzed (Participants) | 157 | 166
Participants
  Number of Participants YES Observed ≥2-point improvement | 84 | 54
  Number of Participants NO Observed ≥2-point improvement | 73 | 112
Statistical Analysis 1: Comparison: Active vs Vehicle; Test type: Other; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 2.34, 95% CI 2-sided [1.47 to 3.72]

2. Primary Outcome: Observed Change in Participant (Vehicle Arm vs SB Gel 15% Arm) Ranked Gravimetric Sweat Production From Baseline to End of Treatment
Description: Individual gravimetric sweat production values were reported as the combined measured weight (mg) of axillary (right+left axillae) sweat production at each visit. Gravimetric sweat production values were rank-transformed.
  Baseline GSP was the median rank of GSP measurements obtained on Visit 2, Visit 3, and Visit 4.
  End of Treatment GSP was the median rank of GSP measurements obtained on Visit 10, Visit 11, and Visit 12.
  The difference in ranked GSP from baseline to end of treatment (ranked GSP at end of treatment [6 weeks] minus ranked GSP at baseline) was used as the outcome value.
Time Frame: as for outcome 1
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Active | Vehicle
Number analyzed (Participants) | 157 | 165
milligrams | -27.88 (94.670) | -7.24 (99.695)
Statistical Analysis 1: Comparison: Active vs Vehicle; Test type: Other; p = 0.0019, ANCOVA; Mean Difference (Net) = -29.71, 95% CI 2-sided [-48.42 to -11.00], Standard Error of Mean 9.543

ADVERSE EVENTS:
Time Frame: 11-15 weeks
Description: A total of 350 participants were randomized into the study, 173 participants to sofpironium bromide gel,15% and 177 participants to vehicle gel (placebo). All except one participant (349 participants total) received at least one dose of study drug. A subject in the vehicle group was withdrawn from the study before receiving any study treatment because the subject did not meet eligibility criteria.
Arm/Group | Active | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/176
Serious Adverse Events (participants affected / at risk) | 1/173 | 0/176
Other Adverse Events (participants affected / at risk) | 58/173 | 6/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=173) | Vehicle (N=176)
SMALL BOWEL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) — SMALL INTESTINAL OBSTRUCTION
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=173) | Vehicle (N=176)
APPLICATION SITE PAIN (General disorders) | 11 | 3
APPLICATION SITE PRURITUS (General disorders) | 11 | 1
APPLICATION SITE DERMATITIS (General disorders) | 10 | 1
APPLICATION SITE ERYTHEMA (General disorders) | 9 | 1
DRY MOUTH (Gastrointestinal disorders) | 20 | 0
MYDRIASIS (Eye disorders) | 13 | 0
VISION BLURRED (Eye disorders) | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement terms prioritized a multi-center publication at the study end. Should such a publication not be completed, an investigator right to individually publish results of his/her study (limited to his/her site data) was included, if for purely scientific or educational purposes; not for any commercial purposes. PI(s) were to submit draft materials to the Sponsor 60 days prior to Investigator release of individual abstract or manuscript. Additional disclosure restrictions and terms applied.

DOCUMENTS (2):
  • Study Protocol (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT03836287/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT03836287/SAP_001.pdf